CLINICAL TRIAL: NCT00604305
Title: A Randomized Single Blind Comparative Study of the Acuity's C-Well Accommodating Intra Occular Lens (AIOL) Against Alcon's Acrysof
Brief Title: Comperative Trial Between an Accommodative Iol and Monofocal Iol
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Company could not supply the accommodating intraocular lenses for the study
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Yaacov Rozenman, Head of eye department, Shaare Zedek Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6666476CTIL; Rozenman-CWPMS001
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: CATARACT SURGERY

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acrysof (Active Comparator): Routine monofocal IOL
  Interventions: Device: Acrysof
- Acuity's AIOL (Active Comparator): Accomodaing IOL
  Interventions: Device: Acuity's AIOL

INTERVENTIONS:
Device: Acrysof — Monofocal IOL
  Arms: Acrysof
Device: Acuity's AIOL — Accommodating IOL
  Arms: Acuity's AIOL

SUMMARY:
a comparison of two intraocular lenses in regard of accommodative power.

DETAILED DESCRIPTION:
A new accommodating IOL (Acuity Ltd, Israel) will be compared with Alcon's Acrysof for 1 year for visual acuity and distance and near best corrected visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30 and 65
* Required cataract operation in one or both eyes
* BCVA potetial at least 20/30
* Clear intraoccular media
* Willing to participate in study as evidenced by signing a written Informed Consent

Exclusion Criteria:Main

* Prior surgery at the selected eye
* No light perception or poor potential for improvement
* Phacodonesis and damaged zonules
* Pupil size at least 6 mm.
* History of uveitis
* Macular disease decreasing vision below 20/30
* Amblyopia
* Axial length shorter than 21 mm and longer than 25 mm

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-03; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
distance and near visual acuity | 1 year

SECONDARY OUTCOMES:
centration pco | 1 year